CLINICAL TRIAL: NCT01509586
Title: A Test of Short and Long Term Naturalistic Outcomes of Smokers Who Sample Smokeless Tobacco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00007428; R01CA154992 (NIH)
Record Dates: First submitted 2011-12-14; First posted 2012-01-13 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Smoking; Smoking Cessation
Keywords: smoking; smoking cessation; Potentially Reduced Exposure Products (PREPs)
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PREP (Potentially Reduced Exposure Product) Group (Experimental)
  Interventions: Drug: Potentially Reduced Exposure Product (PREP): a smokeless, spit-free tobacco product
- cigarette group (No Intervention)

INTERVENTIONS:
Drug: Potentially Reduced Exposure Product (PREP): a smokeless, spit-free tobacco product — The PREP Group will be given a sample supply of a PREP product that is already on the market. It is unclear if it is safer than cigarettes, and that is why it is classified as a Potentially Reduced Exposure Product. It provides both nicotine and tobacco in the form of a pouch that can be thrown away after used. Unlike chewing tobacco, there is no need for spitting with this product. There are multiple flavors and participants will have his/her choice of preferred flavor. This group will be asked to sample the product and use it in several ways, but whether a participant uses the product or not is up him/her.
  Arms: PREP (Potentially Reduced Exposure Product) Group

SUMMARY:
This nationwide telephone and mail- based research study will recruit 1,400 cigarette smokers who are not motivated to quit to test the effects of a marketed oral, non-combustible smokeless tobacco product on cigarette smoking behaviors. It will also track the participants' usage patterns of the smokeless tobacco product.

Half of the participants will receive a new, potentially safer tobacco product during the first six weeks of the study, and half will not. During this six-week period, each participant will complete three brief phone interviews. After this first six week period, participants will complete 6 other brief follow-up interviews, where they will answer questionnaires about their smoking habits.

ELIGIBILITY:
Inclusion Criteria:

* age >=19
* a daily cigarette smoker of >=10 cigs/day
* English speaking
* live in the contiguous U.S.
* unmotivated to quit smoking in the next 30 days

Exclusion Criteria:

* no use of smokeless tobacco in past six months
* not breastfeeding, pregnant, or planning a pregnancy
* devoid of any recent (past 6 months) cardiovascular trauma
* no quit attempt of >=1 week in past 6 months
* no use of pharmacotherapy to quit smoking in past 3 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1236 (Actual)
Dates: Start 2011-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Carpenter, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Carpenter MJ, Wahlquist AE, Burris JL, Gray KM, Garrett-Mayer E, Cummings KM, Alberg AJ. Snus undermines quit attempts but not abstinence: a randomised clinical trial among US smokers. Tob Control. 2017 Mar;26(2):202-209. doi: 10.1136/tobaccocontrol-2015-052783. Epub 2016 Apr 12. PMID 27071730

RESULTS

PARTICIPANT FLOW:
Groups:
- Cigarette Group: This group will smoke their normal cigarettes as much or as little as they want to.
Period: Overall Study
Arm/Group | PREP (Potentially Reduced Exposure Product) Group | Cigarette Group
Started | 626 (Week 0) | 610 (Week 0)
Week 3 | 574 | 585
Week 6 | 551 | 585
Week 10 | 537 | 574
Week 14 | 528 | 566
Week18 | 529 | 555
Week 32 (Month 6) | 504 | 523
Week 46 | 483 | 494
Week 58 (Month 12) | 492 | 499
Completed | 626 (final intent to treat sample) | 610 (final intent to treat sample)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PREP (Potentially Reduced Exposure Product) Group | Cigarette Group | Total
Number analyzed (Participants) | 626 | 610 | 1236
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (12.5) | 48.7 (12.6) | 48.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 438 | 397 | 835
  Male | 188 | 213 | 401
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 557 | 531 | 1088
  African-American | 56 | 61 | 117
  Other | 13 | 18 | 31
Intend to quit smoking, next month [Mean (Standard Deviation); unit: units on a scale] — 0 - 10 scale, where 0 is no intent to quit and 10 is the most intent to quit smoking in the next 30 days
  units on a scale | 1.4 (2.3) | 1.3 (2.4) | 1.4 (2.4)
Confidence to quit smoking [Mean (Standard Deviation); unit: units on a scale] — 0 -10 scale, where 0 is no confidence to quit smoking and 10 is the most confidence to quit smoking, in the next 30 days
  units on a scale | 2.6 (3.1) | 2.7 (3.0) | 2.7 (3.1)
Cigarettes per day [Mean (Standard Deviation); unit: average cigarettes per day at baseline] | 20.1 (8.7) | 19.9 (8.4) | 20.0 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Quit Attempts and Abstinence
Description: % of study participants making a quit attempt or staying abstinent from smoking during the study
  Notes:
  Floating abstinence: Any 7-day period of non-smoking, ever within study. PPA: point-prevalence abstinence
Time Frame: From study enrollment through end of one-year follow up
Measure: Number; unit: percentage of participants
Arm/Group | PREP (Potentially Reduced Exposure Product) Group | Cigarette Group
Number analyzed (Participants) | 626 | 610
percentage of participants
  Any quit attempt, ever within study | 25.7 | 30.8
  Any 24 h quit attempt, ever within study | 19.8 | 25.6
  Floating abstinence | 14.9 | 16.2
  Week 32 PPA | 6.2 | 5.6
  Week 58 PPA | 5.1 | 5.6

ADVERSE EVENTS:
Time Frame: Adverse events were asked to both groups at all 8 follow-up interviews (weeks 3, 6, 10, 14, 18, 32, 46, and 58). Numbers below are cumulative of all adverse events reported at all 8 follow-up interviews.
Arm/Group | PREP (Potentially Reduced Exposure Product) Group | Cigarette Group
Serious Adverse Events (participants affected / at risk) | 3/626 | 3/610
Other Adverse Events (participants affected / at risk) | 458/626 | 414/610
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PREP (Potentially Reduced Exposure Product) Group (N=626) | Cigarette Group (N=610)
Death (General disorders) | 3 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PREP (Potentially Reduced Exposure Product) Group (N=626) | Cigarette Group (N=610)
nausea (Gastrointestinal disorders) | 93 | 82
headache (General disorders) | 79 | 93
heartburn (Gastrointestinal disorders) | 68 | 51
mouth soreness (Gastrointestinal disorders) | 46 | 43
dizziness or lightheadnedness (General disorders) | 54 | 61
dry mouth (General disorders) | 53 | 57
sore jaw (General disorders) | 14 | 18
excessive salivation (General disorders) | 29 | 15
insomnia (General disorders) | 66 | 70
hiccups (Gastrointestinal disorders) | 44 | 21
burning in throat/mouth (Gastrointestinal disorders) | 59 | 21
other (General disorders) | 338 | 332

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No